CLINICAL TRIAL: NCT04526977
Title: Differences in Susceptibility and Cytokine Profile, Specific CD4/CD8 T Cell Response, Toll Like Receptors (TLRs) and Killer Immunoglobulin-like Receptors (KIRs) Among HIV-1-infected Individuals With Previous or Current COVID-19
Brief Title: Differences in Immune Response Among HIV-1-infected Individuals With Previous or Current COVID-19 (CoVIHDis).
Acronym: CoVIHDis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asociacion para el Estudio de las Enfermedades Infecciosas (Network)
Responsible Party: Sponsor
Other Study IDs: EC 273/20
Record Dates: First submitted 2020-08-22; First posted 2020-08-26 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Covid19; Immune Suppression; HIV-1-infection
Keywords: HIV; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: HIV-1 infected individuals with previous or current diagnosis of SARS-CoV-2 infection, defined as the presence of suggestive symptoms and a positive PCR from the nasopharyngeal swab.
  Interventions: Diagnostic Test: Immune response study
- Controls: HIV-1-infected individuals of the same age (range, 5 years) and sex, who not have been diagnosed of clinical (asymptomatic) or confirmed SARS CoV-2 infection, but were positive for IgG antibodies (controls group 1) or with no evidence of SARS-CoV-2 infection (no previous neither current symptoms, negative for IgM/IgG antibodies, controls group 2)
  Interventions: Diagnostic Test: Immune response study

INTERVENTIONS:
Diagnostic Test: Immune response study — * ACE2 and CD26 receptor study
  * Cytokine profile: Quantification of plasma cytokine levels
  * SARS-CoV-2 CD4/CD8 T cell response
  * TLR7/8 activation
  * KIR characterization

SUMMARY:
People living with HIV could have different susceptibility and outcome to the SARS CoV-2 infection. The risk of SARS CoV-2 infection in this population could be no related to HIV infection, immunodepression or antiretroviral therapy, but to the different susceptibility as measured by ACE2 or CD26 receptors. Also, patients with HIV-1 infection could have different cytokine profile and cellular immune response after SARS-CoV-2 infection, leading to a differential outcome,

DETAILED DESCRIPTION:
Since March 2020, the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) pandemic has affected almost five million people in 168 countries on five continents, with more than 300.000 deaths (1-4). The scientific evidence so far does not suggest that people with HIV-1 have an increased risk of serious complications if they develop COVID-19 disease (5-7). In our recent work, we have shown in a few patients that people with HIV-1 under antiretroviral treatment, with undetectable viral load and a CD4 count greater than 200 cells/mm3, do not have a higher risk of developing serious complications than people without HIV-1, but also HIV-1 infected patients does not seem to be protected of the so-called cytokine storm (8-11). Like in the general population, they would be more likely to develop serious complications if they are older and with previous pathologies (comorbidity), such as high blood pressure, diabetes, cardiovascular disease, chronic lung disease, cancer or immunosuppression (congenital, acquired or due to treatment with immunosuppressive drugs). Thus, people with HIV-1 who are immunocompromised with a CD4 count less than 200 cells/mm3, regardless of whether or not they take antiretroviral treatment should be considered among the vulnerable groups and therefore at an increased risk of developing serious clinical complications associated to COVID-19 (12-14). It should be noted, however, that, so far, there is no enough scientific evidence that can confirm this possibility (10,15-17).

Since March 2020, the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) pandemic has affected almost five million people in 168 countries on five continents, with more than 300.000 deaths (1-4). The scientific evidence so far does not suggest that people with HIV-1 have an increased risk of serious complications if they develop COVID-19 disease (5-7). In our recent work, we have shown in a few patients that people with HIV-1 under antiretroviral treatment, with undetectable viral load and a CD4 count greater than 200 cells/mm3, do not have a higher risk of developing serious complications than people without HIV-1, but also HIV-1 infected patients does not seem to be protected of the so-called cytokine storm (8-11). Like in the general population, they would be more likely to develop serious complications if they are older and with previous pathologies (comorbidity), such as high blood pressure, diabetes, cardiovascular disease, chronic lung disease, cancer or immunosuppression (congenital, acquired or due to treatment with immunosuppressive drugs). Thus, people with HIV-1 who are immunocompromised with a CD4 count less than 200 cells/mm3, regardless of whether or not they take antiretroviral treatment should be considered among the vulnerable groups and therefore at an increased risk of developing serious clinical complications associated to COVID-19 (12-14). It should be noted, however, that, so far, there is no enough scientific evidence that can confirm this possibility (10,15-17).

Indeed, there are two main questions for the management of this disease in this population, the real incidence of COVID 19 (susceptibility) and if the immune response could be different in those who were already coinfected.

1. The differences in susceptibility to infection could be related to host factors. Thus, it is important to characterize and genotyping the main receptor for SARS-CoV-2, ACE2, and other related receptor, such as CD26, to explore the genetic background affecting the real incidence of this disease, along CD4 count and antiretroviral therapy.
2. People with HIV-1 have an impaired immune system, especially in those with less than 200 CD4 cells/mm3. Hence, the immune response in these individuals could be weaker than in general population, including the cytokine response reported after SARS-CoV-2 infection (18-20). In addition, the specific CD4/CD8 T cell response could be altered due to the HIV-1 infection and the level of immunosuppression. This specific T cell response could be a good marker for the presence or persistence of immunity against SARS-CoV-2 infections.

In addition, the first line of immune defense is the interaction of the virus with innate immunity cell members. The toll like receptors (TLRs) family is a group of pattern recognition receptors that include many different molecules (21-23). These bindings can activate dendritic cells, monocytes, macrophages. There is an important RNA and DNA connection, activation of TLRs, the production of type I interferons, and the development of some autoimmune diseases. TLR7 and TLR8 specifically recognize simple-chain RNA of viruses and are expressed in endosomal membranes. TLR8 is expressed in regulatory cells (Treg) and its activation results in inhibition of its regulatory functions. Natural killer cells (NK) respond to alterations of class I HLA molecules present in infected cells (24-26). An increase in class I HLA expression could lead to an increase in NK activation by increasing its ability to produce IFN-gamma. Therefore, the reasons for KIR binding are often variable between individuals and between populations. However, there are no data about TLRs activation and KIRs binding in HIV infected patients with SARS CoV-2 infection.

This project is designed to improve scientific knowledge and give answers to the actual clinical questions regarding SARS-CoV-2 infection in people living with HIV-1. It could be of importance to determine the risk of infection not related to HIV-related factors, and to ascertain the adequation of the immune response of HIV infected patients after a SARS-CoV-2, identifying therefore those at risk of severe disease.

ELIGIBILITY:
Inclusion Criteria:

* adult (>18 year-old), confirmed HIV-1-infection, and provide written informed consent, with previous SARS CoV-2 infection as demonstrated by clinical and a positive PCR (cases) or no previous compatible symptoms and no diagnosis of SARS-CoV-2 infection (controls, classified according to serological determination)

Exclusion Criteria:

* unable to provide a written informed consent.
* immunological alterations (chronic intake of corticoid or immunosuppresants)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected patients in regular follow up
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Changes in immune cellular response | 3 months
  Differences in cellular response to SARS-COV-2 peptides

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Casado, PhD, Principal Investigator — Hospital Ramon y Cajal
Locations (1):
- Hospital Ramon y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No